CLINICAL TRIAL: NCT00288301
Title: North Carolina WISEWOMAN Study - Weight-Wise Program
Brief Title: North Carolina WISEWOMAN: Weight-Wise Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency); North Carolina Department of Health and Human Services (Other Government)
Responsible Party: Beverly Garcia, The Unviersity of North Carolina at Chapel Hill
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 00893-05
Record Dates: First submitted 2006-02-06; First posted 2006-02-07 (Estimated); Last update posted 2010-06-10 (Estimated); Status verified 2010-06

CONDITIONS: Overweight; Obesity
Keywords: diet; physical activity; weight management
MeSH Terms: conditions — Overweight; Obesity; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Special Intervention
  Interventions: Behavioral: Weight loss intervention
- 2 (Experimental): Delayed intervention
  Interventions: Behavioral: Weight loss intervention

INTERVENTIONS:
Behavioral: Weight loss intervention — weight loss intervention

SUMMARY:
The purpose of this study is to test the effectiveness of a weight loss and weight loss maintenance intervention among low income women, conducted in a community health center setting.

DETAILED DESCRIPTION:
In the North Carolina WISEWOMAN Project, nearly three-fourths of all participants are either overweight or obese. Through control of weight, cardiovascular disease risk factors such as hypertension, dyslipidemia, and type 2 diabetes can be reduced along with their associated mortality. While there is some evidence of successful weight loss programs in the scientific literature, there are limited data on strategies to improve the weight loss outcomes of African Americans and other lower income populations and how to maintain weight loss over the long term with strategies that are feasible for health care agencies that service primarily lower income populations. We have designed a program to test intervention strategies to improve the weight loss outcomes of the WISEWOMAN population. Specifically, the purpose of the North Carolina WISEWOMAN Weight Control Pilot Study, "Weight-Wise" Program, is to test the effectiveness of a weight loss and weight loss maintenance intervention among WISEWOMAN participants, conducted in a community health center in Wilmington, NC. The Weight-Wise Program was launched in February 2005 and will continue through the Spring of 2007.

The study design and intervention are briefly described. Each WISEWOMAN participant was invited to a screening visit at the health center. During an interview with a research assistant, the participant answered a series of questions about her health history, diet, physical activity, and weight management behaviors, and psycho-social attributes. She also had her height, weight, blood pressure, and body composition measured. A non-fasting venous blood specimen was taken to measure her blood lipids (total and HDL-cholesterol) and random blood glucose. Additional baseline measures for psycho-social variables were obtained via telephone administration. Participants who completed the screening visit, phone interview, and met all eligibility requirements were randomized to two treatment groups: the Special Intervention (SI) group, and the Delayed Intervention (DI) group. Participants assigned to the SI group began the 4-month weight loss phase of the study in April 2005, while DI participants will wait until the end of this first program offering to begin the weight loss program. [DI participants are considered the 'control' group.]

The intervention program, called "Weight-Wise", consists of a four-month weight loss intervention phase, and a one-year maintenance phase. During the weight loss intervention, participants are offered 16 weekly group education sessions taught by a health counselor. The study goal for weight loss during this period is 10 or more pounds. Each session lasts about 120 minutes and includes the following elements: participant weigh-in, group sharing and problem-solving, discussion of a weight control topic (nutrition, physical activity, or behavior change), moderate physical activity and/or taste-testing. Study participants who complete the weight loss program and lose 8 or more pounds will be eligible to continue in the maintenance phase of the intervention. During the 1-year maintenance phase (which will start at the end of the weight loss phase for both SI and DI), participants in the SI group will receive 1 individual face-to-face contact with the health counselor, 8 monthly phone contacts, and 3 group sessions. The DI group will receive 1 individual face-to-face contact and 11 phone contacts from the health counselor during their maintenance intervention. After the weight loss phase and after 6 and 12 months of the maintenance intervention, both SI and DI participants will return to the clinic for follow-up data collection.

ELIGIBILITY:
Inclusion Criteria:

* Women 40-64 years old
* Gross income less than or equal to 200% federal poverty level
* BMI 25-45 inclusive
* Permission of health care provider if present with diabetes or previous CVD event
* English speaking

Exclusion Criteria:

* Medical condition for which weight loss is contraindicated, e.g. malignancy or other serious illness
* CVD event in past 3 months
* Self-reported history of renal disease
* Weight loss greater than 20 lbs in last 3 months
* Any history of gastric bypass surgery, stomach stapling or liposuction
* Planning to leave area before study period ends
* Current participation in another clinical trial
* Pregnant, breastfeeding or planning a pregnancy before the end of the study
* Current use of medications to treat psychosis or manic-depressive illness

Ages: 40 Years to 64 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 151 (Actual)
Dates: Start 2005-02; Primary Completion 2007-05 (Actual); Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
body weight | 4 months

CONTACTS AND LOCATIONS:
Overall Officials: Carmen Samuel-Hodge, PhD, RD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- New Hanover Community Health Center, Wilmington, North Carolina, United States

REFERENCES:
- [Derived] Samuel-Hodge CD, Johnston LF, Gizlice Z, Garcia BA, Lindsley SC, Gold AD, Braxton DF, Keyserling TC. A pilot study comparing two weight loss maintenance interventions among low-income, mid-life women. BMC Public Health. 2013 Jul 15;13:653. doi: 10.1186/1471-2458-13-653. PMID 23855318
- [Derived] Samuel-Hodge CD, Johnston LF, Gizlice Z, Garcia BA, Lindsley SC, Bramble KP, Hardy TE, Ammerman AS, Poindexter PA, Will JC, Keyserling TC. Randomized trial of a behavioral weight loss intervention for low-income women: the Weight Wise Program. Obesity (Silver Spring). 2009 Oct;17(10):1891-9. doi: 10.1038/oby.2009.128. Epub 2009 Apr 30. PMID 19407810